CLINICAL TRIAL: NCT01411267
Title: A Phase I Study of AC220 for Children With Relapsed or Refractory ALL or AML
Brief Title: AC220 for Children With Relapsed/Refractory ALL or AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Ambit Biosciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2009-004
Record Dates: First submitted 2011-08-01; First posted 2011-08-08 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Myelogenous Leukemia, Acute, Childhood
Keywords: Relapse; Lymphoblastic; Leukemia; AC220; Refractory; Myelogenous; Acute; Childhood; Pediatric; ALL; AML
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid; Recurrence; Leukemia | interventions — quizartinib; Cytarabine; Etoposide; etoposide phosphate; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- ALL AC220 @ 25mg/m2/day (Dose Level 1) (Experimental): The starting dose is Dose Level 1 at 25 mg/m2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide; Drug: Methotrexate
- AML AC220 @ 25mg/m2/day (Dose Level 1) (Experimental): The starting dose is Dose Level 1 at 25 mg/m2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide
- ALL AC220 @ 40mg/m2/day (Dose Level 2) (Experimental): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide; Drug: Methotrexate
- ALL AC220 @ 60mg/m2/day (Dose Level 3) (Experimental): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide; Drug: Methotrexate
- ALL AC220 @ 90mg/m2/day (Dose Level 4) (Experimental): If the study dose of 60 mg/m2/day at Dose Level 3 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 4 at 90 mg/m2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 4 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide; Drug: Methotrexate
- ALL AC220 @ 130 mg/m2/day (Dose Level 5) (Experimental): If the study dose of 90 mg/m2/day at Dose Level 4 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 5 at 130 mg/m2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. Dose Level 5 is the highest dose for this study.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide; Drug: Methotrexate
- AML AC220 @ 40mg/m2/day (Dose Level 2) (Experimental): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide
- AML AC220 @ 60mg/m2/day (Dose Level 3) (Experimental): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide
- AML AC220 @ 90mg/m2/day (Dose Level 4) (Experimental): If the study dose of 60 mg/m2/day at Dose Level 3 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 4 at 90 mg/m2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 4 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide
- AML AC220 @ 130mg/m2/day (Dose Level 5) (Experimental): If the study dose of 90 mg/m2/day at Dose Level 4 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 5 at 130 mg/m2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. Dose Level 5 is the highest dose for this study.
  Interventions: Drug: AC220; Drug: Cytarabine; Drug: Etoposide

INTERVENTIONS:
Drug: AC220 — Dose assigned at study entry. AC220 will be given orally once daily on days 7-28.
  Other Names: Quizartinib
Drug: Cytarabine — All patients receive 1000 mg/m2/day IV given every 12 hours on days 1 through 5. Additionally, AML patients and patients with ambiguous leukemia receive cytarabine intrathecally on day "1" of course 1 and 2. Dose defined by age:
  * 20 mg for patients age <1 yr
  * 30 mg for patients age 1-1.99 years of age
  * 50 mg for patients age 2-2.99 years of age
  * 70 mg for patients >3 years of age
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar®-U; Arabinosylcytosine
Drug: Etoposide — 150 mg/m2/day IV on days 1 through 5.
  Other Names: VePesid®; Etopophos; VP-16; Toposar®; Etoposide phosphate
Drug: Methotrexate — IT methotrexate given intrathecally to patients with ALL on day "0" of course 1 and 2. Dose defined by age
  * 6 mg for patients age < 1yr
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Other Names: MTX; Amethopterin; Otrexup™; Rasuvo®; Rheumatrex®; Trexall™; Methotrexate Sodium
  Arms: ALL AC220 @ 130 mg/m2/day (Dose Level 5); ALL AC220 @ 25mg/m2/day (Dose Level 1); ALL AC220 @ 40mg/m2/day (Dose Level 2); ALL AC220 @ 60mg/m2/day (Dose Level 3); ALL AC220 @ 90mg/m2/day (Dose Level 4)

SUMMARY:
This is a phase I study of the investigational drug AC220 combined with cytarabine and etoposide in pediatric patients with relapsed acute lymphoblastic leukemia (ALL) and acute myelogenous leukemia (AML).

DETAILED DESCRIPTION:
This is a study for pediatric patients with relapsed acute lymphoblastic leukemia (ALL) or acute myelogenous leukemia (AML). Some people diagnosed with leukemia have changes in a receptor located on the surface of white blood cells called FLT3. This is known as a FLT3 mutation. FLT3 plays an important role in the way cells grow and divide. In normal cells, the FLT3 receptor is switched off most of the time and only switches on when it gets a chemical signal from outside. But cells with the FLT3 mutation have the grow signal permanently switched on. This means leukemia cells with the FLT3 mutation are growing and dividing all the time. Doctors have found that people with leukemia cells that carry FLT3 mutations are less likely to go into remission with chemotherapy and have a higher risk of the leukemia coming back after treatment.

This is a study of an investigational drug called AC220. AC220 is considered investigational because it has not been approved in the United States by the Food and Drug Administration (FDA). AC220 is a drug which is able to "turn off" the FLT3 grow signal. AC220 will be given with cytarabine and etoposide to treat the relapsed leukemia. This is a phase I study, which means that the study is being done to find the highest dose of AC220 that can be given safely with the drugs cytarabine and etoposide to children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than 1 month and ≤ 21 years of age at study entry.
* Patients must have a diagnosis of relapsed/refractory AML, ALL or acute leukemia of ambiguous lineage and meet the following criteria:

  1. Patients with AML or leukemia with ambiguous lineage must have greater than or equal to 5% blasts in the bone marrow.
  2. Patients with ALL must have an M3 marrow (marrow blasts >25%).
  3. Patients with ALL must have MLL gene rearrangement or hyperdiploid >50 chromosomes.
  4. Patients with treatment related AML (t-AML) are eligible, provided they meet all other eligibility criteria.
* Karnofsky > 50% for patients >16 years of age and Lansky >50% for patients ≤16 years of age.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  * Myelosuppressive chemotherapy:

    * Patients with ALL who relapse during standard maintenance therapy are eligible at time of relapse.
    * For patients with ALL and AML who relapse while they are receiving cytotoxic therapy, at least 14 days must have elapsed since the completion of cytotoxic therapy.
    * Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of AC220.
    * Patients who have received other FLT3 inhibitors (ex. lestaurtinib, sorafenib) are eligible for this study.
  * Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor.
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  * XRT: 2 wks must have elapsed since local palliative XRT for CNS chloromas; No washout period is necessary for other chloromas; at least 3 months must have elapsed if prior TBI, craniospinal XRT.
  * Hematopoetic Stem Cell Transplant: At least 90 days must have elapsed since hematopoietic stem cell transplant (HSCT) and patients must not have active GVHD.
* Patient must have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Patients must have a calculated creatinine clearance or radioisotope GFR ≥70mL/min/1.73m2 or a normal serum creatinine based on age/gender.
  * Total bilirubin <1.5 x ULN for age or normal conjugated bilirubin.
  * Alanine transaminase (ALT) <5 × ULN (unless related to leukemic involvement).
* Patient must have a shortening fraction of ≥ 27% by echocardiogram, OR an ejection fraction of ≥ 50% by radionuclide angiogram.
* Reproductive Function

  * Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.
  * Female patients with infants must agree not to breastfeed their infants while on this study.
  * Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Patients will be excluded if they have CNS 3 disease.
* Patients will be excluded if they have uncontrolled or significant cardiovascular disease, including:

  * A myocardial infarction within 12 months.
  * Uncontrolled angina within 6 months.
  * Diagnosed or suspected congenital long QT syndrome or any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes [TdP]); any history of arrhythmia will be discussed with the Sponsor's Medical Monitor prior to patient's entry into the study.
  * Prolonged QTcF interval on pre-entry ECG (≥450 ms).
  * Any history of second or third degree heart block (may be eligible if the patient currently has a pacemaker).
  * Heart rate < 50/minute on pre-entry ECG.
  * Uncontrolled hypertension.
  * Complete left bundle branch block.
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or TdP.
* Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.
* Patient is receiving or plans to receive concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients who are concurrently receiving CYP3A4 and 5 inhibitors and inducers

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2013-09-12 (Actual); Study Completion 2013-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Cooper, MD, Study Chair — Children's Healthcare of Atlanta, Emory University
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Cooper TM, Cassar J, Eckroth E, Malvar J, Sposto R, Gaynon P, Chang BH, Gore L, August K, Pollard JA, DuBois SG, Silverman LB, Oesterheld J, Gammon G, Magoon D, Annesley C, Brown PA. A Phase I Study of Quizartinib Combined with Chemotherapy in Relapsed Childhood Leukemia: A Therapeutic Advances in Childhood Leukemia & Lymphoma (TACL) Study. Clin Cancer Res. 2016 Aug 15;22(16):4014-22. doi: 10.1158/1078-0432.CCR-15-1998. Epub 2016 Feb 26. PMID 26920889
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- ALL AC220 @ 25mg/m^2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 25mg/m^2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 40mg/m^2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 40mg/m^2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 60mg/m^2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- AML AC220 @ 60mg/m^2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- ALL AC220 @ 90mg/m^2/Day (Dose Level 4): If the study dose of 60 mg/m^2/day at Dose Level 3 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 4 at 90 mg/m2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 4 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- AML AC220 @ 90mg/m^2/Day (Dose Level 4): If the study dose of 60 mg/m^2/day at Dose Level 3 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 4 at 90 mg/m^2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 4 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- ALL AC220 @ 130mg/m^2/Day (Dose Level 5): If the study dose of 90 mg/m^2/day at Dose Level 4 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 5 at 130 mg/m^2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. Dose Level 5 is the highest dose for this study.
- AML AC220 @ 130mg/m^2/Day (Dose Level 5): If the study dose of 90 mg/m^2/day at Dose Level 4 is well tolerated but does not show sufficient AC220 activity, the study may proceed to Dose Level 5 at 130 mg/m^2/day. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. Dose Level 5 is the highest dose for this study.
Period: Overall Study
Arm/Group | ALL AC220 @ 25mg/m^2/Day (Dose Level 1) | AML AC220 @ 25mg/m^2/Day (Dose Level 1) | ALL AC220 @ 40mg/m^2/Day (Dose Level 2) | AML AC220 @ 40mg/m^2/Day (Dose Level 2) | ALL AC220 @ 60mg/m^2/Day (Dose Level 3) | AML AC220 @ 60mg/m^2/Day (Dose Level 3) | ALL AC220 @ 90mg/m^2/Day (Dose Level 4) | AML AC220 @ 90mg/m^2/Day (Dose Level 4) | ALL AC220 @ 130mg/m^2/Day (Dose Level 5) | AML AC220 @ 130mg/m^2/Day (Dose Level 5)
Started | 0 | 3 | 2 | 5 | 2 | 12 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 2 | 4 | 0 | 10 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients with ALL were enrolled into Dose Level 1
Groups:
- ALL AC220 @ 25mg/m2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 25mg/m2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 40mg/m2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 40mg/m2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 60mg/m2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- AML AC220 @ 60mg/m2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- Total: Total of all reporting groups
Arm/Group | ALL AC220 @ 25mg/m2/Day (Dose Level 1) | AML AC220 @ 25mg/m2/Day (Dose Level 1) | ALL AC220 @ 40mg/m2/Day (Dose Level 2) | AML AC220 @ 40mg/m2/Day (Dose Level 2) | ALL AC220 @ 60mg/m2/Day (Dose Level 3) | AML AC220 @ 60mg/m2/Day (Dose Level 3) | Total
Number analyzed (Participants) | 0 | 3 | 2 | 5 | 2 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] |  | 13.1 [1.8 to 21] | 2.8 [.9 to 19] | 13.1 [1.8 to 21] | 2.8 [.9 to 19] | 13.1 [1.8 to 21] | 11.6 [.9 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3 | 1 | 7 | 14
  Male | 0 | 2 | 0 | 2 | 1 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 1 | 4 | 7
  Not Hispanic or Latino | 0 | 2 | 1 | 4 | 1 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 0 | 2 | 2 | 2 | 1 | 8 | 15
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 3
# Patients with Prior HSCT [Count of Participants; unit: Participants] | 0 | 3 | 0 | 2 | 0 | 5 | 10
FLT3/ITD+ (FLT3-internal tandem duplication mutation) [Count of Participants; unit: Participants] | 0 | 2 | 0 | 3 | 0 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Dose of AC220 That is Safe and Biologically Active When Given in Sequential Combination With Ara-C/Etoposide
Description: The incidence of dose limiting toxicity (DLT) will be measured. The maximum tolerated dose will be the highest study dose at which 1 or fewer of six patients experience DLT during cycle 1 of therapy. Plasma inhibitor activity (PIA) will be measured Pre-treatment and on Days 7, 14, 21 and 28 of Course 1. For the MTD to be considered biologically active, we will require that 7 of 9 patients achieve PIA of > 90% at 3 of 4 trough time points.
Time Frame: 4 weeks from therapy start
Population: No patients with ALL were enrolled during Dose Level 1.
Measure: Count of Participants; unit: Participants
Groups:
- ALL AC220 @ 25mg/m^2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 25mg/m^2/Day (Dose Level 1): The starting dose is Dose Level 1 at 25 mg/m2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 40mg/m^2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML AC220 @ 40mg/m^2/Day (Dose Level 2): Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL AC220 @ 60mg/m^2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- AML AC220 @ 60mg/m^2/Day (Dose Level 3): Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
Arm/Group | ALL AC220 @ 25mg/m^2/Day (Dose Level 1) | AML AC220 @ 25mg/m^2/Day (Dose Level 1) | ALL AC220 @ 40mg/m^2/Day (Dose Level 2) | AML AC220 @ 40mg/m^2/Day (Dose Level 2) | ALL AC220 @ 60mg/m^2/Day (Dose Level 3) | AML AC220 @ 60mg/m^2/Day (Dose Level 3)
Number analyzed (Participants) | 0 | 3 | 2 | 5 | 2 | 12
Participants
  patient completed therapy without DLT | 0 | 3 | 1 | 4 | 0 | 8
  patients experienced DLT | 0 | 0 | 1 | 0 | 0 | 1
  patients withdrew or not evaluable | 0 | 0 | 0 | 1 | 2 | 3

2. Secondary Outcome: Disease Response
Description: Possible outcomes are: Complete Remission (CR), Complete Remission without Platelet Recovery (CRp), complete response with incomplete hematologic recovery (CRi), Stable Disease, Progressive Disease, Induction Death, or Relapse
Time Frame: 10 weeks
Population: Five of 22 patients were not evaluable for response per protocol because they were removed from protocol therapy prior to disease assessment without meeting PD criteria
Measure: Count of Participants; unit: Participants
Groups:
- Patients With ALL: Patients with a diagnosis of acute lymphocytic leukemia at study entry
- Patients With AML Having FLT3-WT: Patients with a diagnosis of acute myeloid leukemia with internal tandem duplication (ITD) on exon 14 of the FLT3 gene
- Patients With AML Having FLT3-ITD: Patients with a diagnosis of acute myeloid leukemia having the FLT3 wild-type receptor (FLT3-WT)
Arm/Group | Patients With ALL | Patients With AML Having FLT3-WT | Patients With AML Having FLT3-ITD
Number analyzed (Participants) | 3 | 7 | 7
Participants
  CR | 0 | 1 | 1
  CRi | 0 | 0 | 1
  CRp | 0 | 0 | 1
  SD | 1 | 5 | 4
  PD | 2 | 1 | 0

3. Secondary Outcome: Count of Participants According to Inhibition of FLT3 Phosphorylation
Description: PIA samples will be collected pre-treatment and on Days 7, 14, 21 and 28 of Course 1.
Time Frame: 4 weeks from therapy start
Population: Nineteen of 22 patients had PIA assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Receiving Protocol Therapy: All patients receiving protocol therapy
Arm/Group | Patients Receiving Protocol Therapy
Number analyzed (Participants) | 19
Participants
  100% inhibition | 9
  97-99% inhibition | 9
  94% inhibition | 1

ADVERSE EVENTS:
Time Frame: Adverse events and suspected adverse reactions will be collected and reported on the electronic CRFs beginning with the first dose of study therapy until 30 days following the last dose of study therapy (a period of approximately 90 days).
Description: The definitions of AE and SAE do not differ from the clinicaltrials.gov definitions.
Groups:
- ALL Dose Level 1: The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML Dose Level 1: The starting dose is Dose Level 1 at 25 mg/m^2/day. Dose escalation will proceed from level 1 to 2 to 3, and so on, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL Dose Level 2: Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age.
- AML Dose Level 2: Dose escalation will proceed from level 1 to level 2 for AC220 at 40mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Cytarabine will be given to patients with AML on Day 0, dose assigned by age.
- ALL Dose Level 3: Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Methotrexate will be given to patients with ALL on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
- AML Dose Level 3: Dose escalation will proceed from level 2 to 3 for AC220 at 60mg/m^2/day, assuming the maximum tolerated dose is not exceeded. Patients will received etoposide and cytarabine on Days 1-5, and AC220 on Day 7 through 28. IT Cytarabine will be given to patients with AML on Day 0, dose assigned by age. If toxicity at Dose Level 3 would allow further escalation, but demonstrated sufficient AC220 activity, no further dose escalation will be required.
Arm/Group | ALL Dose Level 1 | AML Dose Level 1 | ALL Dose Level 2 | AML Dose Level 2 | ALL Dose Level 3 | AML Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/3 | 2/2 | 3/5 | 1/2 | 3/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/3 | 1/2 | 3/5 | 0/2 | 4/10
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 2/2 | 5/5 | 2/2 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL Dose Level 1 (N=0) | AML Dose Level 1 (N=3) | ALL Dose Level 2 (N=2) | AML Dose Level 2 (N=5) | ALL Dose Level 3 (N=2) | AML Dose Level 3 (N=10)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest wall pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Not Specified (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Blood infections of non-specified lineage
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin & subcutaneous tissue disorder-Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection and Infestations - Rhinovirus (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - Staphylococcus epidermidis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - streptococcal pharyngitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0)
Infections and Infestations - Pseudomonas (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL Dose Level 1 (N=0) | AML Dose Level 1 (N=3) | ALL Dose Level 2 (N=2) | AML Dose Level 2 (N=5) | ALL Dose Level 3 (N=2) | AML Dose Level 3 (N=10)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (5) | 1 (1) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (6)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 9 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Infections and infestations - Other - Not otherwise Specified (Infections and infestations) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The lineage of the infection was not recorded nor specified
Lung infection (Infections and infestations) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0
Nausea (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (7)
Pain (General disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 7 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin & subcutaneous tissue disorder-Other - Not otherwise specified (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 — The lineage of these skin and subcutaneous tissue disorders were not specified
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
White blood cell decreased (Investigations) | 0 | 3 (4) | 1 (1) | 5 (5) | 1 (1) | 6 (6)
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Perirectal Abcess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pilonidal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Blood Culture infection (Infections and infestations) | 0 | 2 (2) | 1 (1) | 0 | 0 | 1 (2)
Headache (General disorders) | 0 | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachypnea (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhea (General disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0
Erythmea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Irritation to central line site (General disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0
Left neck peeling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Drainage & reddened skin at Hickman CL site (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Ara-C Skin Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Skin Nodules - Not otherwise specified (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Strep Veridans Bacteremia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Rash on Chest and Upper Arms (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days